CLINICAL TRIAL: NCT06532890
Title: Optimal Pediatric Heart Transplant Immunosuppression With MicroRNAs
Acronym: OPTIMA
Status: Recruiting | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: INOVA-2024-197; Enduring Hearts Awards#1248960 (Other: AHA - American Heart Association)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Failure; Graft Rejection
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to discover circulating microRNAs (associated with drug doses and levels) that can be used to characterize the overall immune state in pediatric heart transplant patients and predict patients that will go on to develop infection and rejection. MicroRNAs (miRs) are small, non-coding RNA molecules that regulate gene expression and serve as molecular biomarkers found in the circulation.

DETAILED DESCRIPTION:
The study objectives will be accomplished in a prospective, multicenter observational, longitudinal cohort study that includes 100-150 Pediatric Heart Transplant (PHT) patients from the United States. Patients will be screened for eligibility and enrolled 10-50 days after PHT. Study participation will last 24 months.

All patients will follow the center's standard of care surveillance schedule after transplant. Blood samples will be collected for miR evaluation at:

1. specified time intervals after transplant and
2. when a clinical event of interest occurs, including treated rejection, or infection.

Research samples will be collected and used to evaluate microRNA expression as well as other biomarkers related to heart transplantation and immunosuppression medications. Additional data collection will include demographics, medical history, medications, human leukocyte (HLA)/donor specific antibody (DSA) evaluations, endomyocardial biopsy (EMB), echocardiography, donor-derived cell-free DNA (dd-cfDNA), and other post-transplant events and testing.

This work will form the basis for a non-invasive, genomic blood test that can be used to monitor patients after heart transplant to mitigate complications of over-immunosuppression, such as infection, without increasing the risks of under-immunosuppression, such as rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years at time of transplant listing
* Subject is within 10-50 days post-orthotopic heart transplant at time of enrollment.
* Planned follow-up at the transplant center for a minimum of one-year.
* Caregiver able and willing to comply with the study visit schedule, study procedures, and study requirements.

Exclusion Criteria:

* Recipient of a multi-organ transplant
* History of prior solid organ transplant before the index heart transplant
* Ongoing mechanical circulatory support or hemodynamic instability after transplant
* Active infection requiring either a) hospitalization or b) treatment with antimicrobial drugs (does not include prophylaxis for infection or suppressive antibiotics given after transplant)
* History of treated rejection prior to study enrollment
* Inability to collect specified blood volume after enrollment and prior to 50 days post-transplant

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients ≤ 18 years of age at time of transplant listing from geographically and socioeconomically diverse regions of the U.S. who have undergone orthotopic heart transplant (OHT).
  Patients will be screened for eligibility and enrolled 10-50 days after pediatric heart transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Time-to-Event Analysis of Circulating microRNAs (miRs) Predicting Infection in Pediatric Heart Transplant Recipients | up to 2 years post-transplant
  A time-to-event analysis will be performed to identify specific circulating microRNAs (miRs) that predict the risk of infection in heart transplant recipients. Infections are defined as any bacterial, viral, fungal, or opportunistic infection leading to: 1) hospitalization, 2) prescription of antimicrobial therapy, or 3) reduction in immunosuppression.
Time-to-Event Analysis of Circulating microRNAs (miRs) Predicting Rejection in Pediatric Heart Transplant Recipients | up to 2 years post-transplant
  A time-to-event analysis will be performed to identify specific circulating microRNAs (miRs) that predict the risk of rejection in heart transplant recipients. Rejection is defined as treated rejection based on 1) endomyocardial biopsy (EMB) pathology, 2) unexplained graft dysfunction, or 3) molecular testing; leading to treatment with pulse dose steroids, monoclonal antibodies, plasmapheresis, and/or intravenous immunoglobulin (IVIg).

CONTACTS AND LOCATIONS:
Overall Officials: Palak Shah, MD, Principal Investigator — Inova Schar Heart and Vascular; Jason Goldberg, MD, Study Director — Inova L.J. Murphy Children's Hospital
Locations (7):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Inova Health System, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah P, Agbor-Enoh S, Bagchi P, deFilippi CR, Mercado A, Diao G, Morales DJ, Shah KB, Najjar SS, Feller E, Hsu S, Rodrigo ME, Lewsey SC, Jang MK, Marboe C, Berry GJ, Khush KK, Valantine HA; GRAfT Investigators. Circulating microRNAs in cellular and antibody-mediated heart transplant rejection. J Heart Lung Transplant. 2022 Oct;41(10):1401-1413. doi: 10.1016/j.healun.2022.06.019. Epub 2022 Jun 28. PMID 35872109
- [Background] Shah P, Bristow MR, Port JD. MicroRNAs in Heart Failure, Cardiac Transplantation, and Myocardial Recovery: Biomarkers with Therapeutic Potential. Curr Heart Fail Rep. 2017 Dec;14(6):454-464. doi: 10.1007/s11897-017-0362-8. PMID 28940102